CLINICAL TRIAL: NCT02878057
Title: Multicenter Phase II Study of Apatinib in Patients With HER-2 Negative Advanced Breast Cancer With Chest Wall Metastasis
Brief Title: Multicenter Phase II Study of Apatinib in Patients With Advanced Breast Cancer(CABC006)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Hebei Medical University Fourth Hospital (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); Shanxi Province Cancer Hospital (Other)
Responsible Party: Principal Investigator, Li Huiping, Head of the department of breast oncology, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016YJZ19
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Results first posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
Keywords: Apatinib; HER-2 Negative; Chest wall Metastasis; Multicenter Phase II Study; Breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Advanced Breast Cancer (Experimental): Patients With HER-2 Negative Advanced Breast Cancer With Chest Wall Metastasis; Dosing regimen: apatinib tablets: 500 mg, Po, QD; 4 weeks as a cycle, continuous treatment until disease progression, death or intolerable toxicity (giving endocrine therapy simultaneously if hormone receptor positive)
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Dosing regimen: apatinib tablets: 500 mg, Po, QD; 4 weeks as a cycle, continuous treatment until disease progression, death or intolerable toxicity (giving endocrine therapy simultaneously if hormone receptor positive)
  Other Names: Apatinib Mesylate Tablets

SUMMARY:
The treatment of the patients with recurrent and metastatic breast cancer remains a major problem. There is still a lack of effective targeted therapy for Her-2 negative breast cancer.Based on the present researches on the anti-angiogenesis drugs in advanced breast cancer, the investigators believe that it is necessary to further explore the efficacy and safety of apatinib in advanced breast cancer.

DETAILED DESCRIPTION:
With the comprehensive treatment of breast cancer wildly used in the clinical practice, the life quality of the patients with breast cancer has been improved greatly, and the survival of the patients has been extended as well. However, the treatment of the patients with recurrent and metastatic breast cancer remains a major problem. There is still a lack of effective targeted therapy for Her-2 negative breast cancer.

Based on the present researches on the anti-angiogenesis drugs in advanced breast cancer, the investigators believe that it is necessary to further explore the efficacy and safety of apatinib in advanced breast cancer. The aim of this research is to evaluate the progression-free survival (PFS) of the patients with HER-2 negative advanced breast cancer with chest wall metastasis in the treatment of apatinib.

ELIGIBILITY:
Inclusion Criteria:

1. HER-2 negative advanced breast cancer with chest wall metastasis confirmed by histology or cytological examination (patients who have received anthracyclines and/or paclitaxel in adjuvant chemotherapy).
2. Patients with recurrence or metastasis who have received no more than two lines of chemotherapy.
3. If hormone receptor is positive, endocrine therapy must have been performed for the patients with recurrence or metastasis, or the recurrence or metastasis occurred in less than two years of endocrine therapy.
4. ≥ 18 years old.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
6. A life expectancy of more than 3 months.
7. At least one measurable site of disease confirmed by CT or MRI according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 criteria was required.
8. If the target lesions are lymph nodes, the short diameter is required to be less than 1.5cm and the target lesions are not suitable for surgical treatment; target lesions have not been in radiotherapy or recurred in the radiation field.
9. Baseline blood routine examination in accordance with the following criteria: neutrophil counts more than 1.5*109/L; platelet counts greater than 100*109/L; hemoglobin greater than 9 g/dL (blood transfusion is allowed to achieve or maintain the index)
10. Liver function in accordance with the following criteria: total bilirubin less than 1.5 times the upper limit of normal value; aspartate aminotransferase (AST), alanine aminotransferase (ALT) less than 2.5 times the upper limit of normal value, less than 5 times the upper limit of normal value in patients with liver metastases.
11. Renal function in accordance with the following criteria: serum creatinine less than 1.25 times the upper limit of normal value, or the creatinine clearance rate calculated greater than 50 mL/min;
12. Women with fertility are willing to take contraceptive measures in the trial: when seven days before the drug delivery of serum or urine pregnancy test negative.

Exclusion Criteria:

1. receiving radiation therapy 28 days before enrolled. Radiotherapy before enrollment to relieve the metastatic bone pain is allowed, but medullary bone radiated should not exceed 30% of the total amount;
2. symptomatic central nervous system metastases;
3. current or recent (30 days before enrollment) use of another study drug or being involved in another clinical study;
4. Other malignant tumors that have occurred within 5 years (except for the cured or well-controlled cervical carcinoma in situ, skin squamous cell carcinoma, or skin basal cell carcinoma);
5. With hypertension and the blood pressure cannot be reduced to the normal range through antihypertensive drug treatment (systolic blood pressure greater than or equal to 140 mmHg or diastolic blood pressure greater than or equal to 90 mmHg).
6. With grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTc interval more than or equal to 450 ms for men, more than or equal to 470 ms for female);
7. according to the criteria of NYHA, cardiac insufficiency of grade III and IV or left ventricular ejection fraction (LVEF) less than 50% revealed by echocardiography;
8. abnormal coagulation function (INR > 1.5 or prothrombin time (PT) > ULN+4 seconds or APTT >1.5 times the ULN), with bleeding tendency or under thrombolysis or anticoagulation therapy;
9. within 3 months before enrollment, clinically significant bleeding symptoms occur, or having obvious bleeding tendency, such as gastrointestinal bleeding, bleeding gastric ulcer, occult blood + + and above in baseline period, or suffering from vasculitis, et al;
10. within 4 months before enrollment receiving major surgery or getting severe traumatic injury, fracture or ulcer;
11. having factors that affect the absorption of the oral drugs obviously, such as the inability to swallow, chronic diarrhea and intestinal obstruction, et al;
12. urine routine test with urinary protein more than ++, or 24 hour urinary protein more than 1.0 g;
13. with symptomatic serous cavity effusion, which needs to be surgically managed (including pleural effusion, ascites, pericardial effusion);
14. with other possible conditions that can affect the clinical research or evaluation of the results judged by the researchers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-09-02 (Actual); Study Completion 2020-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huiping Li, MD, Study Chair — Peking University Cancer Hospital & Institute

IPD SHARING:
Plan to Share IPD: Yes
all information will shared with IPD or other researhers
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Dec. 2020
Access Criteria: published journal
URL: https://www.baidu.com/

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Hao Y, Xu J, Murray T, Thun MJ. Cancer statistics, 2008. CA Cancer J Clin. 2008 Mar-Apr;58(2):71-96. doi: 10.3322/CA.2007.0010. Epub 2008 Feb 20. PMID 18287387
- [Background] Weidner N, Semple JP, Welch WR, Folkman J. Tumor angiogenesis and metastasis--correlation in invasive breast carcinoma. N Engl J Med. 1991 Jan 3;324(1):1-8. doi: 10.1056/NEJM199101033240101. PMID 1701519
- [Background] D'Agostino RB Sr. Changing end points in breast-cancer drug approval--the Avastin story. N Engl J Med. 2011 Jul 14;365(2):e2. doi: 10.1056/NEJMp1106984. Epub 2011 Jun 27. No abstract available. PMID 21707384
- [Background] Miller K, Wang M, Gralow J, Dickler M, Cobleigh M, Perez EA, Shenkier T, Cella D, Davidson NE. Paclitaxel plus bevacizumab versus paclitaxel alone for metastatic breast cancer. N Engl J Med. 2007 Dec 27;357(26):2666-76. doi: 10.1056/NEJMoa072113. PMID 18160686
- [Background] Miles DW, Chan A, Dirix LY, Cortes J, Pivot X, Tomczak P, Delozier T, Sohn JH, Provencher L, Puglisi F, Harbeck N, Steger GG, Schneeweiss A, Wardley AM, Chlistalla A, Romieu G. Phase III study of bevacizumab plus docetaxel compared with placebo plus docetaxel for the first-line treatment of human epidermal growth factor receptor 2-negative metastatic breast cancer. J Clin Oncol. 2010 Jul 10;28(20):3239-47. doi: 10.1200/JCO.2008.21.6457. Epub 2010 May 24. PMID 20498403
- [Background] Robert NJ, Dieras V, Glaspy J, Brufsky AM, Bondarenko I, Lipatov ON, Perez EA, Yardley DA, Chan SY, Zhou X, Phan SC, O'Shaughnessy J. RIBBON-1: randomized, double-blind, placebo-controlled, phase III trial of chemotherapy with or without bevacizumab for first-line treatment of human epidermal growth factor receptor 2-negative, locally recurrent or metastatic breast cancer. J Clin Oncol. 2011 Apr 1;29(10):1252-60. doi: 10.1200/JCO.2010.28.0982. Epub 2011 Mar 7. PMID 21383283
- [Background] Valachis A, Polyzos NP, Patsopoulos NA, Georgoulias V, Mavroudis D, Mauri D. Bevacizumab in metastatic breast cancer: a meta-analysis of randomized controlled trials. Breast Cancer Res Treat. 2010 Jul;122(1):1-7. doi: 10.1007/s10549-009-0727-0. Epub 2010 Jan 9. PMID 20063120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: finished recritment
Period: Overall Study
Arm/Group | Advanced Breast Cancer
Started | 30
Completed | 26
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- Advanced Breast Cancer: Patients With HER-2 Negative Advanced Breast Cancer With Chest Wall Metastasis;
  Dosing regimen: apatinib tablets: 500 mg, Po, QD; 4 weeks as a cycle, Apatinib: Dosing regimen: apatinib tablets: 500 mg, Po, QD; 4 weeks as a cycle, continuous treatment until disease progression, death or intolerable toxicity (giving endocrine therapy simultaneously if hormone receptor positive)
Arm/Group | Advanced Breast Cancer
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 49.5 [35 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Lines of Chemotherapy Prior to Enrollment [Count of Participants; unit: Participants]
  1 | 4
  2 | 10
  ≥3 | 16

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: evaluation per 2 cycles (8 weeks), up to 6 months;From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 6 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Advanced Breast Cancer
Number analyzed (Participants) | 26
months | 4.9 [2.1 to 8.3]

2. Primary Outcome: Overall Survival
Description: survival from first dose to death or last follow up
Time Frame: evaluation per 2 cycles (8 weeks), up to 55 months
Population: Patients With HER-2 Negative Advanced Breast Cancer With Chest Wall Metastasis;
Measure: Median (Full Range); unit: months
Arm/Group | Advanced Breast Cancer
Number analyzed (Participants) | 26
months | 18 [3 to 55]

3. Secondary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Objective response rate = CR + PR.
Time Frame: evaluation per 2 cycles (8 weeks), up to 55 months
Population: Patients With HER-2 Negative Advanced Breast Cancer With Chest Wall Metastasis;
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Breast Cancer
Number analyzed (Participants) | 26
Participants | 11

4. Secondary Outcome: Disease Control Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression Disease (PD), >=20% increase in the sum of the longest diameter of target lesions or appearance of new lesions; Stable Disease (SD), between PR and PD.
  Disease control rate (DCR) = CR + PR + SD.
Time Frame: evaluation per 2 cycles (8 weeks), up to 55 months
Population: Patients With HER-2 Negative Advanced Breast Cancer With Chest Wall Metastasis;
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Breast Cancer
Number analyzed (Participants) | 26
Participants | 20

5. Secondary Outcome: Number of Participants With Adverse Events
Description: all kind of adverse events, including hypertension, proteinuria, nausea, fatigue, and bilirubin increase.
Time Frame: evaluation per 2 cycles (8 weeks), up to 55 months
Population: Patients With HER-2 Negative Advanced Breast Cancer With Chest Wall Metastasis
Measure: Count of Participants; unit: Participants
Arm/Group | Advanced Breast Cancer
Number analyzed (Participants) | 30
Participants | 15

ADVERSE EVENTS:
Time Frame: through study completion, an median of 18 months
Description: The apatinib dose given was reduced from 500mg to 250mg for 60% of patients because of side effects.
Arm/Group | Advanced Breast Cancer
All-Cause Mortality (participants affected / at risk) | 2/30
Serious Adverse Events (participants affected / at risk) | 12/30
Other Adverse Events (participants affected / at risk) | 1/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced Breast Cancer (N=30)
proteinuria (Renal and urinary disorders) | 6
Hypertension (Cardiac disorders) | 2
Fatigue (General disorders) | 1
Bilirubin increased (Hepatobiliary disorders) | 2
Transaminase increased (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Advanced Breast Cancer (N=30)
Infection (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/57/NCT02878057/Prot_SAP_000.pdf